CLINICAL TRIAL: NCT06986395
Title: The Efficacy of Blood Flow Restriction Training in Elderly Patients With Sarcopenia.
Brief Title: Blood Flow Restriction Training for Age-Related Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuxiang Liang, Physiotherapist-in-Charge, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241201
Record Dates: First submitted 2025-05-20; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-01

CONDITIONS: Sarcopenia in Elderly
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFRT Group (Experimental): "Blood flow restriction training with 20% 1RM loading, pneumatic cuff pressure 80-100mmHg (arms)
  Interventions: Device: Blood Flow Restriction Training (BFRT)
- CRT Group (Active Comparator): Conventional resistance training at 65-75% 1RM intensity using weights/elastic bands, matched frequency/duration
  Interventions: Other: Conventional Resistance Training (CRT)

INTERVENTIONS:
Device: Blood Flow Restriction Training (BFRT) — Standard progressive resistance exercise at 65-75% 1RM intensity using weights/elastic bands
  Arms: BFRT Group
Other: Conventional Resistance Training (CRT) — Standard progressive resistance exercise at 65-75% 1RM intensity using weights/elastic bands
  Arms: CRT Group

SUMMARY:
Brief Title: Safe Exercise for Age-Related Muscle Loss in Hospitalized Seniors

Summary:

This study compares two exercise methods to help older hospital patients (age 65+) rebuild muscle strength after being diagnosed with sarcopenia (age-related muscle loss). We want to know if using special pressure cuffs during light exercise works better than traditional strength training alone.

Who Can Join:

Hospitalized seniors with stable health conditions Excludes those with severe disabilities, dementia, or certain blood circulation problems

What We'll Do:

40 participants will be randomly assigned to either:

Traditional Training Group:

Uses weights/bands at 65-75% max capacity Arm/leg exercises 3x/week for 4 weeks

Pressure Cuff Training Group:

Uses special cuffs on arms/thighs during lighter exercises (20% max capacity) Same exercise frequency with controlled pressure for safety

What We'll Measure:

Handgrip strength (main test at 0/4/12 weeks) Walking speed, balance tests, quality of life surveys Any side effects like dizziness/nausea

Safety First:

Doctors will check your health before starting. Nurses will monitor every session. We use medical-grade cuffs with safe pressure limits (arm: 80-100mmHg, thigh: 150-200mmHg). You can stop anytime if uncomfortable.

Why This Matters:

This could help hospitalized seniors regain strength faster using gentler exercises. All activities are supervised by rehabilitation specialists at West China Hospital, with ethics committee approval (IRB number required).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged ≥65 years
* Diagnosed with sarcopenia per EWGSOP2019 criteria
* Acute medical conditions stabilized for ≥4 weeks (e.g., resolved infections, controlled heart failure)

Exclusion Criteria:

* Severe disability (Barthel Index ≤40)
* Significant cognitive impairment (MMSE ≤18) or major psychiatric disorders (DSM-5 criteria)
* Contraindications to blood flow restriction training:

  * History/predisposition to deep vein thrombosis
  * Coagulopathy (INR >1.5, platelets <100×10⁹/L)
  * Symptomatic varicose veins (CEAP class C4-C6)
  * Uncontrolled hypertension (BP >160/100 mmHg)
  * Chronic lymphedema (ISL stage II-III)
  * Peripheral artery disease (ABI ≤0.7)
  * Active systemic infection (CRP >10 mg/L)
  * Malignancy (except non-melanoma skin cancer)
  * Severe renal impairment (eGFR <30 mL/min/1.73m²)
  * Acute coronary syndrome within 3 months

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in Handgrip Strength | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 12)

SECONDARY OUTCOMES:
6-Meter Walking Speed | Baseline (Week 0), Follow-up (Week 12)
Short Physical Performance Battery (SPPB) | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 12)
Timed Up and Go Test (TUG) | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 12)
MBI | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 12)

IPD SHARING:
Plan to Share IPD: Undecided